CLINICAL TRIAL: NCT00041119
Title: Cyclophosphamide And Doxorubicin (CA) (4 VS 6 Cycles) Versus Paclitaxel (4 VS 6 Cycles) As Adjuvant Therapy For Breast Cancer in Women With 0-3 Positive Axillary Lymph Nodes:A 2X2 Factorial Phase III Randomized Study
Brief Title: Four Versus Six Cycles of Cyclophosphamide/Doxorubicin or Paclitaxel in Adjuvant Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-40101; CDR0000069444 (Registry Identifier: PDQ (Physician Data Query)); NCI-2009-00474 (Registry Identifier: CTRP (Clinical Trials Reporting System)); U10CA180821 (NIH); NCT00698217 (obsolete NCT alias)
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: stage IB breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (CA for 4 courses) (Active Comparator): Patients receive cyclophosphamide IV and doxorubicin hydrochloride IV on day 1. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: AC regimen; Drug: doxorubicin hydrochloride
- Arm II (CA for 6 courses [closed to accrual 12/15/2007]) (Experimental): Patients receive cyclophosphamide IV and doxorubicin hydrochloride IV on day 1. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: AC regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride
- Arm III (paclitaxel for 4 courses) (Experimental): Patients receive paclitaxel IV over 3 hours on day 1. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: AC regimen; Drug: paclitaxel
- Arm IV (paclitaxel for 6 courses [closed 12/15/2007]) (Experimental): Patients receive paclitaxel IV over 3 hours on day 1. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: AC regimen; Drug: paclitaxel

INTERVENTIONS:
Drug: AC regimen — Given IV
Drug: cyclophosphamide — Given IV
  Arms: Arm II (CA for 6 courses [closed to accrual 12/15/2007])
Drug: doxorubicin hydrochloride — Given IV
  Arms: Arm I (CA for 4 courses); Arm II (CA for 6 courses [closed to accrual 12/15/2007])
Drug: paclitaxel — Given IV
  Arms: Arm III (paclitaxel for 4 courses); Arm IV (paclitaxel for 6 courses [closed 12/15/2007])

SUMMARY:
This randomized phase III trial studies cyclophosphamide and doxorubicin hydrochloride compared with paclitaxel as adjuvant therapy in treating breast cancer in women with 0-3 positive axillary lymph nodes. Giving additional cancer treatment after surgery may help to lower the risk that the cancer will come back (adjuvant therapy). Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin hydrochloride, and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether the standard adjuvant therapy of cyclophosphamide and doxorubicin hydrochloride is more effective than paclitaxel in treating women with breast cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the equivalence of paclitaxel given every two weeks with cyclophosphamide and doxorubicin hydrochloride (CA) given every two weeks as adjuvant therapy for women with 0-3 positive axillary lymph nodes, for disease-free survival.

II. To determine if longer therapy, 12 weeks, is superior to shorter therapy, 8 weeks, of either CA or paclitaxel for disease-free survival for women with primary breast cancer with 0-3 positive axillary lymph nodes.

SECONDARY OBJECTIVES:

I. To determine the equivalence of paclitaxel given every two weeks with CA given every two weeks, and the potential superiority of longer vs. shorter therapy, in relation to overall survival, local control (regardless of metastatic status) and time to distant metastases (regardless of local recurrence status).

II. To compare toxicities of short and long course CA and paclitaxel as adjuvant therapy for women with 0-3 positive axillary lymph node breast cancer.

III. To determine the effect of long and short course CA and paclitaxel on the induction of menopause for pre-menopausal patients.

IV. To assess the discrepancy of myelosuppression among the common multidrug resistance protein 1 (MDR1) haplotypes in the CA treatment arm.

V. To assess the effect of MDR1 haplotypes on disease-free survival (DFS) adjusted for treatment.

VI. Exploratory analysis of the effect of cytochrome P450, family 3, subfamily A, polypeptide 5 (CYP3A5), cytochrome P450, family 2, subfamily C, polypeptide 8 (CYP2C8), and cytochrome P450, family 2, subfamily B, polypeptide 6 (CYP2B6) polymorphisms on DFS and toxicity.

VII. To identify genetic markers associated with the risk of developing neutropenia in adriamycin/ cyclophosphamide-treated breast cancer patients.

VIII. To identify genetic markers associated with the risk of developing peripheral neuropathy in paclitaxel-treated breast cancer patients.

IX. To identify genetic markers associated with differences in the efficacy of each chemotherapy regimen.

X. To examine genetic associations with other response and toxicity phenotypes that become apparent during future analysis of Cancer and Leukemia Group B (CALGB) 40101 data.

XI. To identify copy number variants associated with adriamycin/cyclophosphamide-induced neutropenia and paclitaxel-induced peripheral neuropathy.

OUTLINE: Patients are randomized to 1 of 4 treatment arms.

ARM I: Patients receive cyclophosphamide intravenously (IV) and doxorubicin hydrochloride IV on day 1. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive cyclophosphamide IV and doxorubicin hydrochloride IV on day 1. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.

ARM III: Patients receive paclitaxel IV over 3 hours on day 1. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity.

ARM IV: Patients receive paclitaxel IV over 3 hours on day 1. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Note: Randomization to Arms II and IV is no longer available, effective 12/15/2007.

After completion of study treatment patients are followed up for 4-6 weeks, every 6 months for 2 years, and then annually for up to 13 years.

ELIGIBILITY:
Eligibility Criteria:

* Patients must have histologically confirmed invasive carcinoma of the female breast, with 0-3 positive axillary lymph nodes
* Patients must have 0-3 positive axillary lymph nodes to be eligible for this study; patients with node-negative breast cancer should have sufficiently "high risk" disease to warrant chemotherapy; as general guidelines, node-negative patients with tumors of >= 1 cm or estrogen or progesterone receptor negative tumors of any size may be eligible; ultimately though, the definition of "high risk" may be determined by the treating physician, and if the treating physician feels the patient warrants chemotherapy, the patient is eligible; for patients with 1-3 positive axillary nodes, the patient is eligible regardless of primary breast tumor characteristics, if in the opinion of the treating physician, chemotherapy is deemed potentially beneficial to the patient
* If the patient has had a negative sentinel node biopsy, then no further axillary dissection is required, and the patient is determined to be node-negative; if an axillary dissection, without a sentinel node biopsy, is performed to determine nodal status, at least six axillary lymph nodes must be removed and analyzed and negative for the patient to be considered node-negative; axillary nodes with single cells or tumor clusters =< 0.2 mm by either hematoxylin and eosin stain (H&E) or immunohistochemistry (IHC), will be considered node-negative; lymph nodes positive for polymerase chain reaction (PCR) with tumor cells/clusters =< 0.2 mm will be considered node-negative; any axillary lymph node with tumor clusters > 0.2 mm will be considered positive
* If the patient has a sentinel node biopsy and one of the sentinel nodes is positive, as defined by tumor clusters > 0.2 mm, an axillary dissection must be performed; a total of at least 6 axillary lymph nodes, including sentinel nodes plus the subsequent dissection, must be removed for the patient to be eligible; of all the lymph nodes removed from both the sentinel node procedure and the axillary dissection, 1-3 must be positive for the patient to be eligible as a node-positive patient; if an axillary dissection is done without a sentinel node procedure, at least 6 lymph nodes must be removed and a 1-3 nodes must be positive for the patient to be considered node-positive and eligible for this study
* Determination of involvement of axillary nodes with metastatic cancer will follow the revised tumor-node-metastasis (TNM) staging system: axillary nodes with single cells with tumor clusters =< 0.2 mm, by either H&E or immunohistochemistry (IHC), will be considered negative axillary node; lymph nodes positive for PCR with tumor cells/clusters < 0.2 mm will be considered negative axillary node; any axillary lymph node with clusters > 0.2 mm will be considered to be positive
* Patients with estrogen-receptor and/or progesterone receptor negative, positive, or unknown tumors are eligible; estrogen-receptor (ER) and progesterone receptor (PgR) assays should be performed by immunohistochemical methods according to the local institution's standard protocol
* Patients with human epidermal growth factor receptor 2 (HER2) positive, negative or unknown disease are eligible for this trial; patients whose tumors are HER2 positive by either immunohistochemistry 3+ staining or demonstrate gene amplification by fluorescence in situ hybridization (FISH) may receive trastuzumab
* There must be negative tumor margins for invasive cancer and ductal carcinoma in situ (DCIS) in the case of mastectomy or lumpectomy; lobular carcinoma in situ (LCIS) is acceptable at the margin
* Patients with multi-centric breast cancer are eligible as long as all known disease is resected with negative margins, and have 0-3 positive axillary lymph nodes
* Patients must be registered within 84 days of the last breast surgery; patients must have undergone either modified radical mastectomy or lumpectomy; for patients undergoing sentinel node sampling or axillary dissection a simple mastectomy is acceptable; lumpectomy patients must receive radiation therapy; for patients treated with radiation therapy prior to chemotherapy, the patients should be registered on this study after the conclusion of radiation, with chemotherapy administration beginning within 7 days of registration

  * All primary breast and axillary node surgery must be completed prior to enrollment on study
* No previous trastuzumab, chemotherapy or hormonal therapy for this malignancy, except for tamoxifen therapy
* No previous anthracycline chemotherapy for any disease
* Patients with locally advanced breast cancer, inflammatory breast cancer or metastatic breast cancer are not eligible; patients with involvement of dermal lymphatics on pathology are not eligible, even if there are no clinical signs of inflammatory cancer
* Patients with bilateral, synchronous invasive breast cancer are eligible as long as both primary tumors; if a patient has an invasive cancer on one side that meets the eligibility criteria, and DCIS or LCIS on the contralateral side, the patient is eligible; DCIS or LCIS should be managed according to institutional guidelines
* Patients must be disease free from prior malignancies for > 5 years, except for curatively treated basal cell or squamous cell carcinoma of the skin or carcinoma-in-situ of the cervix; patients with a history of invasive breast cancer, or DCIS are eligible if they have been disease free for > 5 years; patients with a history of LCIS are eligible regardless of the interval from diagnosis
* Common Toxicity Criteria (CTC) performance status 0-1
* Women must not be pregnant or nursing
* Concomitant exogenous hormone therapy, including oral contraceptives, post-menopausal hormone replacement therapy, and raloxifene must be stopped before patients can be enrolled
* Patients may have received up to 4 weeks of tamoxifen therapy for this malignancy and still be eligible for this study; patients who received tamoxifen or another selective estrogen receptor modulator (SERM) for prevention or for other indicators (e.g. osteoporosis) are eligible; tamoxifen therapy or other SERMs must be discontinued before the patient is enrolled on this study

  * The use of bisphosphonates for the treatment of osteoporosis is permitted; the use of raloxifene is not permitted are enrollment on this study
* Patients must have adequate organ function including no active congestive heart failure, and no myocardial infarction < 6 months from time of registration
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Platelet count >= 100,00/mm^3
* Creatinine =< 2.0 mg/dl
* Bilirubin =< 1.5 x upper limits of institutional normal
* Patients may be enrolled on adjuvant bisphosphonate studies; patients may be enrolled concurrently or sequentially on 40101 and bisphosphonate trials
* Patients may be enrolled on adjuvant hormonal studies approved by CALGB or Cancer Trials Support Unit (CTSU), such as the Suppression of Ovarian Function Trial (SOFT) and Tamoxifen and Exemestane Trial (TEXT) trials

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3871 (Actual)
Dates: Start 2002-05; Primary Completion 2012-04 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence N. Shulman, MD, Study Chair — Dana-Farber Cancer Institute
Locations (527):
- United States (526):
  - Regional Medical Center, Anniston, Alabama
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Valley Medical Oncology, Fremont, California
  - Washington Township Hospital, Fremont, California
  - California Cancer Center - Woodward Park Office, Fresno, California
  - Cancer Care Associates, Fresno, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Valley Care Medical Center, Pleasanton, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - Mercy Regional Cancer Center at Mercy Medical Center, Redding, California
  - University of California Davis Cancer Center, Sacramento, California
  - Naval Medical Center - San Diego, San Diego, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Sutter Health - Western Division Cancer Research Group, San Rafael, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Memorial Hospital Cancer Center - Colorado Springs, Colorado Springs, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Herbert D. Kerman Regional Oncology Center - Daytona Beach, Daytona Beach, Florida
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Center for Cancer Care and Research at Watson Clinic, LLP, Lakeland, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Integrated Community Oncology Network - Orange Park, Orange Park, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Palm Beach Cancer Institute - West Palm Beach, West Palm Beach, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Alexian Brothers Radiation Oncology, Elk Grove Village, Illinois
  - St. Francis Hospital, Evanston, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Saint James Hospital and Health Centers Comprehensive Cancer Institute - Olympia Fields, Olympia Fields, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Center for Cancer Care at OSF Saint Anthony Medical Center, Rockford, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Heartland Oncology and Hematology, Council Bluffs, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Cancer Resource Center at King's Daughters Medical Center, Ashland, Kentucky
  - Pennington Cancer Center at Baton Rouge General, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - Ochsner Health Center - Covington, Covington, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton MD, Maryland
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Caritas Norwood Hospital, Norwood, Massachusetts
  - NSMC Cancer Center - Peabody, Peabody, Massachusetts
  - Berkshire Hematology Oncology, PC, Pittsfield, Massachusetts
  - Noble Hospital, Westfield, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls Medical Group, PA, Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Hattiesburg Clinic, PA at Forrest General, Hattiesburg, Mississippi
  - Hematology & Oncology Clinic, Hattiesburg, Mississippi
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Skaggs Cancer Center at Skaggs Regional Medical Center, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - St. John's Regional Medical Center, Joplin, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Saint Francis Cancer Treatment Center at Saint Francis Memorial Health Center, Grand Island, Nebraska
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - Callahan Cancer Center at Great Plains Regional Medical Center, North Platte, Nebraska
  - CCOP Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Dana-Farber Cancer Institute at Londonderry, Londonderry, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - UMDNJ University Hospital, Newark, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Mount Sinai Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Fitzpatrick Cancer Center at Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Highland Hospital of Rochester, Rochester, New York
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Faxton Regional Cancer Center, Utica, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Alamance Cancer Center at Alamance Regional Medical Center, Burlington, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Medical Center Cancer Center, Fayetteville, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Maria Parham Medical Center, Henderson, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Granville Medical Center, Oxford, North Carolina
  - Duke Health Raleigh Hospital, Raleigh, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Person Memorial Hospital, Roxboro, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Marion L. Shepard Cancer Center at Beaufort County Hospital, Washington, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Trinity CancerCare Center, Minot, North Dakota
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Cleo Craig Cancer Research Clinic, Lawton, Oklahoma
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Dubs Cancer Center at Rogue Valley Medical Center, Medford, Oregon
  - Providence Cancer Center at PMCC, Medford, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - St. Joseph Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Kent County Memorial Hospital, Warwick, Rhode Island
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Oncology Services of Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Nashville Oncology Associates, PC, Nashville, Tennessee
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Martha Jefferson Hospital Cancer Care Center, Charlottesville, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Virginia Oncology Associates - Hampton, Hampton, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Virginia Cancer Institute - West End, Richmond, Virginia
  - Carilion Cancer Center of Western Virginia, Roanoke, Virginia
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center, Spokane, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Providence Cancer Center at Holy Family Hospital, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Luther Midlelfort Hospital, Eau Claire, Wisconsin
  - Midelfort Clinic - Luther, Eau Claire, Wisconsin
  - Vince Lombardi Cancer Center at Aurora Lakeland Medical Center - Elkhorn, Elkhorn, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercy Regional Cancer Center, Janesville, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Dean Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Marinette, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Columbia-Saint Mary's Cancer Care Center, Milwaukee, Wisconsin
  - Medical Consultants, Limited, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic - Sheboygan, Sheboygan, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Aurora Medical Center, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic - Two Rivers, Two Rivers, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Baldwin RM, Owzar K, Zembutsu H, Chhibber A, Kubo M, Jiang C, Watson D, Eclov RJ, Mefford J, McLeod HL, Friedman PN, Hudis CA, Winer EP, Jorgenson EM, Witte JS, Shulman LN, Nakamura Y, Ratain MJ, Kroetz DL. A genome-wide association study identifies novel loci for paclitaxel-induced sensory peripheral neuropathy in CALGB 40101. Clin Cancer Res. 2012 Sep 15;18(18):5099-109. doi: 10.1158/1078-0432.CCR-12-1590. Epub 2012 Jul 27. PMID 22843789
- [Result] Shulman LN, Cirrincione CT, Berry DA, Becker HP, Perez EA, O'Regan R, Martino S, Atkins JN, Mayer E, Schneider CJ, Kimmick G, Norton L, Muss H, Winer EP, Hudis C. Six cycles of doxorubicin and cyclophosphamide or Paclitaxel are not superior to four cycles as adjuvant chemotherapy for breast cancer in women with zero to three positive axillary nodes: Cancer and Leukemia Group B 40101. J Clin Oncol. 2012 Nov 20;30(33):4071-6. doi: 10.1200/JCO.2011.40.6405. Epub 2012 Jul 23. PMID 22826271
- [Derived] Barginear M, Dueck AC, Allred JB, Bunnell C, Cohen HJ, Freedman RA, Hurria A, Kimmick G, Le-Rademacher JG, Lichtman S, Muss HB, Shulman LN, Copur MS, Biggs D, Ramaswamy B, Lafky JM, Jatoi A. Age and the Risk of Paclitaxel-Induced Neuropathy in Women with Early-Stage Breast Cancer (Alliance A151411): Results from 1,881 Patients from Cancer and Leukemia Group B (CALGB) 40101. Oncologist. 2019 May;24(5):617-623. doi: 10.1634/theoncologist.2018-0298. Epub 2018 Nov 8. PMID 30409792
- [Derived] Shulman LN, Berry DA, Cirrincione CT, Becker HP, Perez EA, O'Regan R, Martino S, Shapiro CL, Schneider CJ, Kimmick G, Burstein HJ, Norton L, Muss H, Hudis CA, Winer EP. Comparison of doxorubicin and cyclophosphamide versus single-agent paclitaxel as adjuvant therapy for breast cancer in women with 0 to 3 positive axillary nodes: CALGB 40101 (Alliance). J Clin Oncol. 2014 Aug 1;32(22):2311-7. doi: 10.1200/JCO.2013.53.7142. Epub 2014 Jun 16. PMID 24934787

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (CA for 4 Courses) | Arm II (CA for 6 Courses [Closed to Accrual 12/15/2007]) | Arm III (Paclitaxel for 4 Courses) | Arm IV (Paclitaxel for 6 Courses [Closed 12/15/2007])
Started | 1142 | 789 | 1151 | 789
Completed | 1142 | 789 | 1151 | 789
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients that were eligible and treated for the study were evaluated
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (CA for 4 Courses) | Arm II (CA for 6 Courses [Closed to Accrual 12/15/2007]) | Arm III (Paclitaxel for 4 Courses) | Arm IV (Paclitaxel for 6 Courses [Closed 12/15/2007]) | Total
Number analyzed (Participants) | 1142 | 789 | 1151 | 789 | 3871
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 978 | 719 | 987 | 715 | 3399
  >=65 years | 164 | 70 | 164 | 74 | 472
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (9.9) | 52.6 (9.1) | 54.0 (9.9) | 52.7 (9.2) | 53.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1142 | 789 | 1151 | 789 | 3871
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Relapse Free Survival (RFS) 4 vs. 6 Cycles
Description: To determine if longer therapy, 12 weeks, is superior to shorter therapy, 8 weeks, of either CA or paclitaxel for relapse-free survival for women with primary breast cancer with 0-3 positive axillary lymph nodes. An assessment of the superiority of 6 cycles over 4 cycles will be conducted. This analysis combines Arm I and Arm III together, and Arm II and Arm IV together.
Time Frame: from baseline up to 4 years
Population: All patients that were eligible and received treatment were analyzed. 700 patients were not included due to the timing that the analysis was performed.
Measure: Median (Full Range); unit: years
Groups:
- 4 Cycles (Arm I and Arm III Combined): Patients receive cyclophosphamide IV and doxorubicin hydrochloride IV OR paclitaxel over 3 hours on day 1. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity.
- 6 Cycles (Arm II and Arm IV Combined): Patients receive cyclophosphamide IV and doxorubicin hydrochloride IV OR paclitaxel over 3 hours on day 1. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | 4 Cycles (Arm I and Arm III Combined) | 6 Cycles (Arm II and Arm IV Combined)
Number analyzed (Participants) | 1593 | 1578
years | NA [NA to NA] — The median has not been reached | NA [NA to NA] — The median has not been reached
Statistical Analysis 1: Comparison: 4 Cycles (Arm I and Arm III Combined) vs 6 Cycles (Arm II and Arm IV Combined); The null hypothesis is that the hazards of both 6 and 4 cycle regimens are equal. The alternative hypothesis is a hazard ratio of 0.77, corresponding to a decrease of 23% in hazard due to longer duration of chemotherapy; Test type: Superiority — If the 5-year DFS for 4 cycles is 84.7% then a decrease of 23% in hazard rate for 6 cycles corresponds to an increase in 5-year DFS to 88%. Assuming a 2-sided significance level of 0.05, there is 90.9% power to detect such an increase at the final analysis conducted 6.4 years after study activation; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.84 to 1.28]

2. Primary Outcome: Duration of Disease Free Survival (RFS)
Description: To determine the equivalence of paclitaxel to CA as adjuvant therapy for women with 0-3 positive axillary lymph nodes, for disease-free survival. Objective progression is defined as the appearance of local (chest wall, axillary, supraclavicular nodes) or distant metastases. The trial is designed to show the equivalence of the experimental agent T with the standard agent combination CA, thus the 4 and 6 course arms of each drug will be combined to conduct this analysis.
Time Frame: from baseline up to 6.4 years
Population: All eligible patients were treated and analyzed.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm V (Arm I and Arm II Combined): Patients receive cyclophosphamide IV and doxorubicin hydrochloride IV on day 1. Treatment repeats every 14 days for 4 or 6 courses in the absence of disease progression or unacceptable toxicity.
- Arm VI (Arm III and Arm IV) Combined: Patients receive paclitaxel IV over 3 hours on day 1. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm V (Arm I and Arm II Combined) | Arm VI (Arm III and Arm IV) Combined
Number analyzed (Participants) | 1931 | 1940
months | NA [NA to NA] — The median for disease free survival was never reached | NA [NA to NA] — The median for disease free survival was never reached
Statistical Analysis 1: Comparison: Arm V (Arm I and Arm II Combined) vs Arm VI (Arm III and Arm IV) Combined; Test type: Equivalence — For T to be considered equivalent to the standard CA, a confidence interval of the hazard ratio of T to CA should be wholly to the left of 1.3, corresponding to a 30% increase in hazard rate. If the 5-year DFS for CA is 88% then an increase of 30% in hazard rate for T corresponds to 5-year DFS of 84.7%. The null hypothesis is that the hazard ratio of T to CA exceeds 1.3. The alternative hypothesis is that the two hazard rates are equivalent; Hazard Ratio (HR) = 1.26, 95% CI 1-sided [upper limit 1.48]

3. Secondary Outcome: Overall Survival (OS)
Description: To determine the equivalence of paclitaxel to CA as adjuvant therapy for women with 0-3 positive axillary lymph nodes, for overall survival. OS will be measured from study entry until death due to any cause. Survivors will be censored at the date of last follow-up.. The trial is designed to show the equivalence of the experimental agent T with the standard agent combination CA, thus the 4 and 6 course arms of each drug will be combined to conduct this analysis.
Time Frame: from baseline up to 5 years
Population: All patients that were eligible and treated for the study were evaluated.
Measure: Number; unit: percentage of participants at 5 years
Groups:
- Cyclophosphamide and Doxorubicin Hydrochloride: Patients receive cyclophosphamide IV and doxorubicin hydrochloride IV on day 1. Treatment repeats every 14 days for 4 or 6 courses in the absence of disease progression or unacceptable toxicity.
- Paclitaxel: Patients receive paclitaxel IV over 3 hours on day 1. Treatment repeats every 14 days for 4 or 6 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Cyclophosphamide and Doxorubicin Hydrochloride | Paclitaxel
Number analyzed (Participants) | 1931 | 1940
percentage of participants at 5 years | 95 | 94
Statistical Analysis 1: Comparison: Cyclophosphamide and Doxorubicin Hydrochloride vs Paclitaxel; Test type: Non-Inferiority or Equivalence — Power calculations were designed to detect effects in the marginal distributions of the two study factors, agent and length, and assume no interaction between the two factors. Calculations also assume exponential DFS and a total of 4556 treated patients accrued over 29 months and followed for four years after accrual termination for a total study time of 6.4 years. We assume the 5-year DFS of CA therapy is 88% and 84.7% for T. These assumptions are based upon results of SWOG 8897; Hazard Ratio (HR) = 1.27, 95% CI 1-sided [upper limit 1.56]

4. Secondary Outcome: Adverse Events
Description: To compare toxicities of short course CA and paclitaxel with long course CA and paclitaxel as adjuvant therapy for women with 0-3 positive axillary lymph node breast cancer. The percentage of patients that received a grade 3 or higher hematologic event will be reported here. We will be combining arm I with arm III, as well as arm II with arm IV. For a complete list of adverse events, please refer to the adverse events section.
Time Frame: from baseline up to 6 weeks post-treatment
Population: 3754 patients were considered evaluable for toxicity that occurred during treatment.
Measure: Number; unit: percentage of patients
Groups:
- 6 Cycles: Patients will either receive cyclophosphamide and doxorubicin hydrochloride for 6 cycles or Paclitaxel for 6 cycles
- 4 Cycles: Patients will either receive cyclophosphamide and doxorubicin hydrochloride for 4 cycles or Paclitaxel for 4 cycles
Arm/Group | 6 Cycles | 4 Cycles
Number analyzed (Participants) | 1528 | 2226
percentage of patients | 38 | 29

5. Secondary Outcome: Time to Distant Metastases
Description: Local control and distant metastasis will be calculated as the cumulative incidence of first local relapse and first distant metastasis, respectively.
Time Frame: from baseline up to 15 years
Population: All patients that were eligible and received treatment were analyzed.
Measure: Median (Full Range); unit: years
Arm/Group | Cyclophosphamide and Doxorubicin Hydrochloride | Paclitaxel
Number analyzed (Participants) | 1931 | 1940
years | NA [NA to NA] — The median has not been reached | NA [NA to NA] — The median has not been reached

6. Secondary Outcome: Local Control
Description: Local control will be calculated as the cumulative incidence of first local relapse.
Time Frame: from baseline up to 15 years
Population: All patients that were eligible and received treatment were analyzed.
Measure: Median (Full Range); unit: years
Arm/Group | Cyclophosphamide and Doxorubicin Hydrochloride | Paclitaxel
Number analyzed (Participants) | 1931 | 1940
years | NA [NA to NA] — The median has not been reached. | NA [NA to NA] — The median has not been reached.

7. Secondary Outcome: Overall Survival (OS) for 4 vs. 6 Cycles
Description: To determine if longer therapy, 12 weeks, is superior to shorter therapy, 8 weeks, of either CA or paclitaxel for overall survival for women with primary breast cancer with 0-3 positive axillary lymph nodes. An assessment of the superiority of 6 cycles over 4 cycles will be conducted. This analysis combines Arm I and Arm III together, and Arm II and Arm IV together.
Time Frame: from baseline up to 4 years
Population: All patients that were eligible and received treatment were analyzed.
Measure: Number; unit: percentage of patients at 4 years
Arm/Group | 6 Cycles | 4 Cycles
Number analyzed (Participants) | 1578 | 2293
percentage of patients at 4 years | 90.9 | 91.8
Statistical Analysis 1: Comparison: 6 Cycles vs 4 Cycles; Test type: Non-Inferiority or Equivalence — Power calculations were designed to detect effects in the marginal distributions of the two study factors, agent and length, and assume no interaction between the two factors. Calculations also assume exponential DFS and a total of 4556 treated patients accrued over 29 months and followed for four years after accrual termination for a total study time of 6.4 years; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [.84 to 1.49]

ADVERSE EVENTS:
Arm/Group | Arm I (CA for 4 Courses) | Arm II (CA for 6 Courses [Closed to Accrual 12/15/2007]) | Arm III (Paclitaxel for 4 Courses) | Arm IV (Paclitaxel for 6 Courses [Closed 12/15/2007])
Serious Adverse Events (participants affected / at risk) | 113/1142 | 104/789 | 59/1151 | 53/789
Other Adverse Events (participants affected / at risk) | 940/1110 | 687/765 | 975/1118 | 668/762
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm I (CA for 4 Courses) (N=1142) | Arm II (CA for 6 Courses [Closed to Accrual 12/15/2007]) (N=789) | Arm III (Paclitaxel for 4 Courses) (N=1151) | Arm IV (Paclitaxel for 6 Courses [Closed 12/15/2007]) (N=789)
Blood disorder (Blood and lymphatic system disorders) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 30/1110 (35) | 29/765 (33) | 1/1118 (1) | 0/762 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 81/1110 (112) | 64/765 (88) | 29/1118 (34) | 19/762 (21)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 3/1110 (4) | 5/765 (6) | 2/1118 (2) | 1/762 (1)
Arrhythmia (Cardiac disorders) | 6/1110 (6) | 5/765 (6) | 7/1118 (8) | 2/762 (4)
Atrial fibrillation (Cardiac disorders) | 1/1110 (1) | 0/765 (0) | 0/1118 (0) | 0/762 (0)
Cardiac disorder (Cardiac disorders) | 1/1110 (1) | 0/765 (0) | 1/1118 (1) | 1/762 (1)
Cardiac pain (Cardiac disorders) | 1/1110 (1) | 0/765 (0) | 0/1118 (0) | 0/762 (0)
Edema (Cardiac disorders) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Left ventricular failure (Cardiac disorders) | 1/1110 (1) | 5/765 (5) | 1/1118 (1) | 0/762 (0)
Myocardial ischemia (Cardiac disorders) | 2/1110 (2) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Vertigo (Ear and labyrinth disorders) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Photophobia (Eye disorders) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Vision blurred (Eye disorders) | 1/1110 (1) | 0/765 (0) | 0/1118 (0) | 0/762 (0)
Abdominal pain (Gastrointestinal disorders) | 1/1110 (2) | 0/765 (0) | 4/1118 (5) | 1/762 (1)
Colitis (Gastrointestinal disorders) | 2/1110 (2) | 2/765 (2) | 1/1118 (1) | 0/762 (0)
Constipation (Gastrointestinal disorders) | 1/1110 (1) | 0/765 (0) | 0/1118 (0) | 0/762 (0)
Diarrhea (Gastrointestinal disorders) | 27/1110 (32) | 24/765 (27) | 11/1118 (11) | 5/762 (5)
Dyspepsia (Gastrointestinal disorders) | 1/1110 (1) | 0/765 (0) | 0/1118 (0) | 0/762 (0)
Dysphagia (Gastrointestinal disorders) | 0/1110 (0) | 2/765 (2) | 0/1118 (0) | 0/762 (0)
Esophagitis (Gastrointestinal disorders) | 4/1110 (4) | 0/765 (0) | 0/1118 (0) | 0/762 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0/1110 (0) | 0/765 (0) | 1/1118 (1) | 0/762 (0)
Gastric ulcer (Gastrointestinal disorders) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 2/762 (2)
Melena/GI bleeding (Gastrointestinal disorders) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Mucositis oral (Gastrointestinal disorders) | 39/1110 (61) | 30/765 (43) | 7/1118 (9) | 4/762 (4)
Nausea (Gastrointestinal disorders) | 12/1110 (15) | 8/765 (9) | 7/1118 (8) | 3/762 (3)
Pancreatitis (Gastrointestinal disorders) | 0/1110 (0) | 2/765 (2) | 0/1118 (0) | 0/762 (0)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1/1110 (1) | 0/765 (0) | 0/1118 (0) | 0/762 (0)
Rectal pain (Gastrointestinal disorders) | 2/1110 (2) | 0/765 (0) | 0/1118 (0) | 0/762 (0)
Typhlitis (Gastrointestinal disorders) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Vomiting (Gastrointestinal disorders) | 7/1110 (8) | 9/765 (10) | 5/1118 (6) | 1/762 (1)
Chest pain (General disorders) | 3/1110 (3) | 2/765 (2) | 1/1118 (1) | 3/762 (3)
Chills (General disorders) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Fatigue (General disorders) | 14/1110 (16) | 12/765 (13) | 4/1118 (5) | 6/762 (6)
Fever (General disorders) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 2/762 (2)
Gait abnormal (General disorders) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Pain (General disorders) | 3/1110 (4) | 2/765 (2) | 0/1118 (0) | 4/762 (4)
Hypersensitivity (Immune system disorders) | 1/1110 (1) | 2/765 (2) | 4/1118 (4) | 6/762 (7)
Catheter related infection (Infections and infestations) | 1/1110 (1) | 1/765 (1) | 2/1118 (2) | 1/762 (1)
Eye infection intraocular (Infections and infestations) | 1/1110 (1) | 0/765 (0) | 0/1118 (0) | 0/762 (0)
Infection (Infections and infestations) | 1/1110 (1) | 0/765 (0) | 0/1118 (0) | 0/762 (0)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 10/1110 (10) | 8/765 (8) | 0/1118 (0) | 0/762 (0)
Infection with unknown ANC (Infections and infestations) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Infection without neutropenia (Infections and infestations) | 7/1110 (8) | 5/765 (5) | 7/1118 (7) | 3/762 (3)
Infectious colitis (Infections and infestations) | 1/1110 (1) | 0/765 (0) | 0/1118 (0) | 0/762 (0)
Peripheral nerve infection (Infections and infestations) | 1/1110 (1) | 0/765 (0) | 0/1118 (0) | 0/762 (0)
Skin infection (Infections and infestations) | 2/1110 (2) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Soft tissue infection (Infections and infestations) | 1/1110 (1) | 0/765 (0) | 0/1118 (0) | 0/762 (0)
Tooth infection (Infections and infestations) | 1/1110 (1) | 0/765 (0) | 0/1118 (0) | 0/762 (0)
Urinary tract infection (Infections and infestations) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Wound infection (Infections and infestations) | 1/1110 (1) | 0/765 (0) | 1/1118 (1) | 0/762 (0)
Wound-infectious (Infections and infestations) | 2/1110 (2) | 3/765 (3) | 0/1118 (0) | 0/762 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0/1110 (0) | 0/765 (0) | 1/1118 (1) | 0/762 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1/1110 (1) | 0/765 (0) | 0/1118 (0) | 0/762 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0/1110 (0) | 1/765 (1) | 1/1118 (2) | 1/762 (1)
Alanine aminotransferase increased (Investigations) | 0/1110 (0) | 1/765 (1) | 1/1118 (1) | 4/762 (4)
Alkaline phosphatase (Investigations) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Amylase increased (Investigations) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Aspartate aminotransferase increased (Investigations) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 2/762 (2)
Blood bilirubin increased (Investigations) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Cardiac troponin T increased (Investigations) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Creatinine increased (Investigations) | 1/1110 (1) | 1/765 (1) | 1/1118 (1) | 0/762 (0)
Fibrinogen for leukemia studies (Investigations) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
INR increased (Investigations) | 1/1110 (2) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Laboratory test abnormal (Investigations) | 1/1110 (1) | 0/765 (0) | 0/1118 (0) | 0/762 (0)
Leukocyte count decreased (Investigations) | 67/1110 (90) | 66/765 (105) | 8/1118 (10) | 2/762 (2)
Lipase increased (Investigations) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Lymphocyte count decreased (Investigations) | 4/1110 (4) | 4/765 (7) | 1/1118 (1) | 1/762 (1)
Neutrophil count decreased (Investigations) | 66/1110 (87) | 61/765 (98) | 10/1118 (11) | 4/762 (4)
Platelet count decreased (Investigations) | 40/1110 (51) | 36/765 (51) | 3/1118 (5) | 5/762 (6)
Anorexia (Metabolism and nutrition disorders) | 5/1110 (5) | 3/765 (3) | 1/1118 (2) | 0/762 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 4/1110 (5) | 2/765 (2) | 4/1118 (6) | 5/762 (6)
Dehydration (Metabolism and nutrition disorders) | 12/1110 (13) | 8/765 (8) | 3/1118 (3) | 2/762 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 0/1110 (0) | 1/765 (1) | 1/1118 (1) | 0/762 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 8/1110 (9) | 2/765 (2) | 1/1118 (2) | 0/762 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1/1110 (1) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/1110 (1) | 0/765 (0) | 1/1118 (1) | 5/762 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0/1110 (0) | 1/765 (1) | 3/1118 (3) | 0/762 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0/1110 (0) | 1/765 (1) | 4/1118 (4) | 5/762 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0/1110 (0) | 0/765 (0) | 1/1118 (1) | 0/762 (0)
Arachnoiditis (Nervous system disorders) | 1/1110 (1) | 0/765 (0) | 0/1118 (0) | 0/762 (0)
Ataxia (Nervous system disorders) | 0/1110 (0) | 0/765 (0) | 1/1118 (1) | 0/762 (0)
Depressed level of consciousness (Nervous system disorders) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Dizziness (Nervous system disorders) | 1/1110 (1) | 1/765 (1) | 0/1118 (0) | 1/762 (1)
Dysgeusia (Nervous system disorders) | 2/1110 (2) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Headache (Nervous system disorders) | 4/1110 (4) | 1/765 (1) | 0/1118 (0) | 4/762 (4)
Ischemia cerebrovascular (Nervous system disorders) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Memory impairment (Nervous system disorders) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Neuralgia (Nervous system disorders) | 1/1110 (2) | 0/765 (0) | 1/1118 (1) | 0/762 (0)
Peripheral motor neuropathy (Nervous system disorders) | 3/1110 (4) | 0/765 (0) | 4/1118 (6) | 7/762 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 9/1110 (10) | 6/765 (7) | 23/1118 (27) | 25/762 (26)
Syncope (Nervous system disorders) | 3/1110 (4) | 2/765 (2) | 0/1118 (0) | 4/762 (4)
Tremor (Nervous system disorders) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Vasovagal episode (Nervous system disorders) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 2/762 (2)
Anxiety (Psychiatric disorders) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Confusion (Psychiatric disorders) | 1/1110 (1) | 1/765 (1) | 0/1118 (0) | 1/762 (1)
Depression (Psychiatric disorders) | 1/1110 (1) | 1/765 (1) | 1/1118 (1) | 1/762 (1)
Hallucinations (Psychiatric disorders) | 1/1110 (1) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Insomnia (Psychiatric disorders) | 1/1110 (1) | 0/765 (0) | 0/1118 (0) | 0/762 (0)
Personality change (Psychiatric disorders) | 0/1110 (0) | 1/765 (1) | 1/1118 (1) | 0/762 (0)
Dysuria (painful urination) (Renal and urinary disorders) | 0/1110 (0) | 1/765 (1) | 1/1118 (1) | 0/762 (0)
Renal failure (Renal and urinary disorders) | 0/1110 (0) | 0/765 (0) | 1/1118 (1) | 0/762 (0)
Urogenital disorder (Renal and urinary disorders) | 1/1110 (1) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Reproductive tract disorder (Reproductive system and breast disorders) | 0/1110 (0) | 0/765 (0) | 1/1118 (1) | 0/762 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1/1110 (1) | 0/765 (0) | 1/1118 (1) | 1/762 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0/1110 (0) | 0/765 (0) | 1/1118 (1) | 1/762 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2/1110 (2) | 2/765 (2) | 0/1118 (0) | 0/762 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3/1110 (3) | 1/765 (1) | 1/1118 (1) | 0/762 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5/1110 (5) | 5/765 (5) | 1/1118 (1) | 3/762 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1/1110 (1) | 2/765 (2) | 1/1118 (1) | 3/762 (3)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2/1110 (2) | 7/765 (7) | 0/1118 (0) | 1/762 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1/1110 (1) | 2/765 (2) | 0/1118 (0) | 0/762 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3/1110 (5) | 1/765 (1) | 3/1118 (3) | 1/762 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 2/1110 (2) | 3/765 (3) | 0/1118 (0) | 0/762 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0/1110 (0) | 0/765 (0) | 1/1118 (1) | 0/762 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0/1110 (0) | 0/765 (0) | 1/1118 (1) | 0/762 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 2/1110 (2) | 0/765 (0) | 1/1118 (1) | 0/762 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0/1110 (0) | 1/765 (1) | 0/1118 (0) | 0/762 (0)
Capillary leak syndrome (Vascular disorders) | 0/1110 (0) | 0/765 (0) | 1/1118 (1) | 0/762 (0)
Hematoma (Vascular disorders) | 0/1110 (0) | 0/765 (0) | 1/1118 (1) | 0/762 (0)
Hemorrhage (Vascular disorders) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Vascular disorders) | 0/1110 (0) | 0/765 (0) | 0/1118 (0) | 1/762 (1)
Hypertension (Vascular disorders) | 0/1110 (0) | 0/765 (0) | 3/1118 (3) | 1/762 (1)
Hypotension (Vascular disorders) | 3/1110 (3) | 3/765 (3) | 0/1118 (0) | 2/762 (2)
Thrombosis (Vascular disorders) | 8/1110 (8) | 7/765 (7) | 6/1118 (6) | 4/762 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (CA for 4 Courses) (N=1110) | Arm II (CA for 6 Courses [Closed to Accrual 12/15/2007]) (N=765) | Arm III (Paclitaxel for 4 Courses) (N=1118) | Arm IV (Paclitaxel for 6 Courses [Closed 12/15/2007]) (N=762)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 44 (52) | 33 (41) | 3 (3) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 698 (1742) | 519 (1789) | 440 (990) | 337 (1034)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphatic disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lymphatics (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transfusion: Platelets (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 2 (2) | 8 (13) | 0 (0) | 2 (3)
Arrhythmia (Cardiac disorders) | 35 (53) | 32 (49) | 39 (57) | 23 (33)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema (Cardiac disorders) | 0 (0) | 5 (5) | 4 (6) | 9 (16)
Left ventricular failure (Cardiac disorders) | 20 (32) | 13 (19) | 26 (47) | 22 (55)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (2)
Eye disorder (Eye disorders) | 3 (3) | 3 (5) | 1 (1) | 1 (2)
Flashing vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 3 (6) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 3 (4) | 4 (7) | 4 (4) | 0 (0)
Watering eyes (Eye disorders) | 4 (5) | 3 (4) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (9) | 2 (2) | 10 (11) | 6 (6)
Anal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 23 (35) | 19 (26) | 13 (14) | 15 (21)
Diarrhea (Gastrointestinal disorders) | 235 (374) | 196 (328) | 241 (349) | 177 (340)
Dry mouth (Gastrointestinal disorders) | 2 (3) | 2 (5) | 3 (3) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 10 (15) | 7 (9) | 3 (4) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 9 (9) | 5 (7) | 0 (0) | 2 (4)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (4) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melena/GI bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 368 (639) | 318 (705) | 132 (179) | 115 (189)
Nausea (Gastrointestinal disorders) | 79 (140) | 67 (126) | 25 (35) | 20 (34)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT studies, if specified in (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 54 (70) | 32 (41) | 6 (6) | 4 (4)
Chest pain (General disorders) | 3 (3) | 4 (4) | 3 (3) | 2 (3)
Chills (General disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Dysmenorrhea (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 73 (137) | 78 (155) | 55 (93) | 52 (100)
Fever (General disorders) | 2 (3) | 2 (2) | 3 (4) | 2 (2)
General symptom (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 2 (2) | 2 (3) | 3 (5) | 0 (0)
Pain (General disorders) | 9 (12) | 8 (12) | 10 (11) | 11 (12)
Hepatic hemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 12 (20) | 10 (13) | 107 (149) | 63 (98)
Immune system disorder (Immune system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 5 (5) | 1 (1) | 1 (1) | 1 (1)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 7 (7) | 12 (12) | 0 (0) | 1 (2)
Infection with unknown ANC (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Infection without neutropenia (Infections and infestations) | 17 (19) | 15 (15) | 14 (15) | 8 (8)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 2 (4) | 1 (1) | 1 (2) | 1 (1)
Wound-infectious (Infections and infestations) | 1 (1) | 2 (4) | 2 (2) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 2 (2) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 10 (10) | 7 (7) | 25 (28) | 14 (21)
Alkaline phosphatase (Investigations) | 4 (4) | 5 (8) | 10 (16) | 11 (22)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 5 (8) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 7 (7) | 13 (17) | 7 (14)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 4 (6)
Coagulopathy (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 2 (4) | 4 (8) | 4 (4) | 3 (3)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (4) | 2 (5) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1) | 2 (4) | 2 (4) | 0 (0)
Leukocyte count decreased (Investigations) | 426 (845) | 358 (929) | 199 (319) | 143 (289)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 21 (26) | 9 (13) | 8 (12) | 3 (3)
Neutrophil count decreased (Investigations) | 353 (683) | 309 (774) | 145 (207) | 115 (198)
Platelet count decreased (Investigations) | 205 (360) | 169 (379) | 125 (209) | 91 (161)
Weight gain (Investigations) | 2 (2) | 4 (5) | 1 (1) | 2 (2)
Weight loss (Investigations) | 4 (5) | 1 (1) | 1 (1) | 0 (0)
Leukopenia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 11 (13) | 8 (12) | 5 (9) | 4 (8)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (5)
Blood glucose increased (Metabolism and nutrition disorders) | 33 (61) | 26 (55) | 57 (101) | 40 (85)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 12 (16) | 2 (3) | 1 (1) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 5 (8) | 2 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 3 (4) | 3 (4) | 3 (3) | 2 (2)
Serum glucose decreased (Metabolism and nutrition disorders) | 2 (2) | 4 (5) | 1 (1) | 2 (5)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 13 (21) | 9 (15) | 8 (8) | 7 (10)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 5 (5)
Serum sodium decreased (Metabolism and nutrition disorders) | 5 (8) | 3 (3) | 5 (6) | 7 (15)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (3) | 3 (5) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 8 (11) | 46 (68) | 37 (64)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 8 (10) | 52 (68) | 25 (37)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 9 (12) | 52 (73) | 49 (82)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 6 (12) | 2 (2)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (5) | 2 (2) | 9 (10) | 2 (2)
Dysgeusia (Nervous system disorders) | 4 (5) | 4 (12) | 7 (8) | 6 (13)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Headache (Nervous system disorders) | 19 (25) | 19 (26) | 14 (19) | 12 (18)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 7 (11)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 17 (20) | 19 (22) | 110 (166) | 108 (221)
Peripheral sensory neuropathy (Nervous system disorders) | 95 (153) | 101 (182) | 650 (1621) | 513 (1786)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sense of smell (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 2 (2) | 5 (5) | 5 (5)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vasovagal episode (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuro-Sensory (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 6 (7) | 5 (6) | 6 (11) | 10 (11)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 6 (7) | 4 (4) | 7 (10) | 8 (15)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 10 (13) | 7 (12) | 8 (10) | 7 (10)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (painful urination) (Renal and urinary disorders) | 1 (2) | 3 (3) | 1 (1) | 3 (3)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urethral hemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 4 (4) | 2 (2) | 2 (2)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 6 (8) | 5 (11) | 3 (3) | 5 (6)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reproductive tract disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Vaginal mucositis (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 5 (10) | 2 (2) | 3 (3)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 10 (15) | 1 (1) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (2) | 2 (2) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 12 (17) | 9 (10) | 8 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 5 (5) | 4 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (5) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 43 (89) | 44 (90) | 37 (64) | 40 (81)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (5)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (11) | 0 (0) | 2 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (3) | 4 (6) | 4 (4) | 3 (6)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (6) | 7 (11) | 6 (11)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 5 (6) | 4 (4) | 14 (20) | 17 (24)
Rash/dermatitis associated with high-dose chemotherapy or BMT studies. (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (4) | 4 (8)
Sweating (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (7) | 2 (3) | 2 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 2 (6) | 3 (8)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 15 (20) | 11 (21) | 17 (27) | 9 (12)
Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 10 (15) | 8 (12)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Phlebitis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 10 (11) | 12 (26) | 3 (4) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less